CLINICAL TRIAL: NCT01917799
Title: Low Dose Aspirin and Low-molecular-weight Heparin in the Treatment of Pregnant Libyan Women With Recurrent Miscarriage
Brief Title: Aspirin, Heparin and Miscarriage
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Khartoum (Other)
Responsible Party: Principal Investigator, Ishag Adam, Professor, University of Khartoum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LDA and LMWH
Record Dates: First submitted 2013-07-31; First posted 2013-08-07 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Pregnancy; Miscarriage
Keywords: Aspirin; Heparin; pregnancy; miscarriage
MeSH Terms: conditions — Abortion, Spontaneous | interventions — Aspirin; Heparin; Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aspirin (Experimental): 75mg tab of aspirin once daily
  Interventions: Drug: Aspirin
- Aspirin + heparin (Active Comparator): 75mg tab of aspirin once daily + 0.4 mL/day of injection of low molecular weight heparin
  Interventions: Drug: Aspirin; Drug: Heparin

INTERVENTIONS:
Drug: Aspirin — 75mg tab of LDA once daily for 7 months
  Other Names: LDA
Drug: Heparin — 0.4 mL/day of the Enoxaparin
  Other Names: Enoxaparin
  Arms: Aspirin + heparin

SUMMARY:
Efficacy of low dose aspirin (LDA) versus LDA plus low-molecular-weight-heparin (LMWH) in patients with a history of recurrent miscarriages.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* History of 2 or more of miscarriage

Exclusion Criteria:

* Twins

Ages: 15 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2009-01; Primary Completion 2013-11 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Number of miscarriages | 3 months
  To compare number of miscarriages between the two groups

CONTACTS AND LOCATIONS:
Locations (1):
- Misurata Teaching Hospital, Misratah, Misurata, Libya

REFERENCES:
- [Derived] Elmahashi MO, Elbareg AM, Essadi FM, Ashur BM, Adam I. Low dose aspirin and low-molecular-weight heparin in the treatment of pregnant Libyan women with recurrent miscarriage. BMC Res Notes. 2014 Jan 9;7:23. doi: 10.1186/1756-0500-7-23. PMID 24405979